CLINICAL TRIAL: NCT02878863
Title: Paeoniflorin Combination of Hepatoprotective Drugs Versus Hepatoprotective Drugs Only for Treatment of Auto-immune Hepatitis
Brief Title: Paeoniflorin Combination of Hepatoprotective Drugs Versus Hepatoprotective Drugs Only for Auto-immune Hepatitis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Xiaoli Fan (Other)
Responsible Party: Sponsor-Investigator, Xiaoli Fan, Principal Investigator, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIH-1
Record Dates: First submitted 2016-08-09; First posted 2016-08-25 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Hepatitis, Autoimmune
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — peoniflorin; Phosphatidylcholines; Silymarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paeoniflorin + phosphatidylcholine or silymarin (Experimental): Paeoniflorin tablets(600mg, tid)combination of phosphatidylcholine or silymarin
  Interventions: Drug: Paeoniflorin + phosphatidylcholine or silymarin
- Phosphatidylcholine or silymarin (Active Comparator): Phosphatidylcholine or silymarin
  Interventions: Drug: Phosphatidylcholine or silymarin

INTERVENTIONS:
Drug: Paeoniflorin + phosphatidylcholine or silymarin
  Other Names: total glucosides of paeony(TGP)+ phosphatidylcholine or silymarin
  Arms: Paeoniflorin + phosphatidylcholine or silymarin
Drug: Phosphatidylcholine or silymarin
  Arms: Phosphatidylcholine or silymarin

SUMMARY:
An open-label,prospective, randomized pilot study to evaluate the efficacy, safety and tolerability of paeoniflorin, for the treatment of autoimmune hepatitis (AIH) with mild necroinflammatory activity on liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-70 years;
* Diagnosed with AIH or primary biliary cirrhosis-autoimmune hepatitis overlap syndrome based on liver biopsy results and without indication of immunosuppressive therapy;
* High levels of alanine aminotransferase (ALT) or aspartate aminotransferase (AST)(1-3 X ULN);
* High levels of IgG(1-1.5 X ULN);
* Liver biopsy showed mild lymphocytic piecemeal necrosis (interface hepatitis);
* Agreed to participate in the trial, and assigned informed consent.

Exclusion Criteria:

* The presence of hepatitis A, B, C, D, or E virus infection;
* Patients with presence of liver cirrhosis or portal hypertension;
* Patients with presence of fulminant liver failure;
* Primary sclerosing cholangitis, non-alcoholic steatohepatitis, drug induced liver disease or Wilson disease confirmed by liver biopsy;
* Pregnant and breeding women;
* Severe disorders of other vital organs, such as severe heart failure, cancer;
* Parenteral administration of blood or blood products within 6 months before screening;
* Recent treatment with drugs having known liver toxicity;
* Taken part in other clinic trials within 6 months before screening.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-03 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Percent of patients that achieve biochemical remission of AIH | Month 6 during treatment with paeoniflorin combination of hepatoprotective drugs or hepatoprotective drugs only
  Biochemical remission is defined as alanine transaminase(ALT),aspartate transaminase(AST) and immunoglobulin G(IgG) within normal limits

SECONDARY OUTCOMES:
Alanine transaminase (ALT) | Month 1, 3, 6
Aspartate transaminase(AST) | Month 1, 3, 6
Immunoglobulin G(IgG) | Month 1, 3, 6
Globin(GLB) | Month 1, 3, 6
Total bilirubin(TB) | Month 1, 3, 6
Direct bilirubin(DB) | Month 1, 3, 6

CONTACTS AND LOCATIONS:
Overall Officials: Li Yang, MD, Study Chair — West China Hospital,Chengdu, Sichuan, China
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided